CLINICAL TRIAL: NCT05659316
Title: New MRI Measurement of Patellar Height in Knee Extension - IES-EV Control Study
Status: Completed | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: RGDS-2019-12-064
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Knee Injuries
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy volunteers: Healthy volunteers without any patellar injury
  Interventions: Other: MRI imaging

INTERVENTIONS:
Other: MRI imaging — Knee MRI imaging

SUMMARY:
The measurement of the patellar height is essential to decide and quantify the surgical correction to be made. The classic index is that of Cato and Deschamps. It has the advantage of its simplicity, with the measurement on a simple profile radiograph of the ratio between the distance from the patella to the tibia and the length of the patella. However, it has the disadvantage of measuring this height in relation to the tibia when the dislocation is located at the level of the patello-trochlear joint. The MRI index of sagittal patellar engagement on the trochlea (IES), described in 2012, does not have this drawback but it does not appear to be reliable: its value depends, in fact, on the flexion of the knee. This flexion, required by the MRI, is variable and is not specified by the radiologist. It is due to the use of an "antenna" that surrounds and lifts the knee.

The hypothesis of the study is that it is possible to determine and validate a new IES, in knee extension and therefore reproducible, thanks to the measurement of knee flexion on MRI. The precise value of this flexion can allow a virtual correction of the original IES to obtain, by mathematical calculation, the new IES in virtual extension.

DETAILED DESCRIPTION:
Patellar instability, usually manifested by recurrent patellar dislocations, is a complex multifactorial pathology. Its treatment associates surgical gestures chosen according to a precise evaluation of the factors of the instability. Five factors are decisive, varying from one subject to another: rupture of the medial patellofemoral ligament, dysplasia of the trochlea, excessive lateralization of the anterior tibial tuberosity (ATT), external torsion of the ATT and patella alta, object of this study. The patella, when it is alta, is an important factor of instability because it is abnormally located above the trochlea in extension of the knee and is no longer guided at the start of flexion: it risks not engaging in the trochlear rail and thus to dislocate at the start of flexion.

The measurement of the patellar height is essential to decide and quantify the surgical correction to be made. The classic index is that of Cato and Deschamps. It has the advantage of its simplicity, with the measurement on a simple profile radiograph of the ratio between the distance from the patella to the tibia and the length of the patella. However, it has the disadvantage of measuring this height in relation to the tibia when the dislocation is located at the level of the patello-trochlear joint. The MRI index of sagittal patellar engagement on the trochlea (IES), described in 2012, does not have this drawback but it does not appear to be reliable: its value depends, in fact, on the flexion of the knee. This flexion, required by the MRI, is variable and is not specified by the radiologist. It is due to the use of an "antenna" that surrounds and lifts the knee.

The hypothesis of the study is that it is possible to determine and validate a new IES, in knee extension and therefore reproducible, thanks to the measurement of knee flexion on MRI. The precise value of this flexion can allow a virtual correction of the original IES to obtain, by mathematical calculation, the new IES in virtual extension.

ELIGIBILITY:
Inclusion Criteria:

* Subject, male or female, over 18 years old
* Subject with an MRI
* Subject without patellar pathology, in particular without patellar instability
* Subject having been informed and not objecting to the use of his data

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subject with knee MRI
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Index of sagittal engagement of the patella (IES) | 1 day
  Measurement of a MRI index of sagittal engagement of the patella (IES) in knee extension at 0°

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé d'Antony, Antony, France

IPD SHARING:
Plan to Share IPD: No